CLINICAL TRIAL: NCT02736422
Title: Assessment of New Magnetic Resonance Imaging (MRI) Pulse Sequences for Imaging Hyperpolarised Xenon in Lung, Heart and Brain in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH15603
Record Dates: First submitted 2016-03-18; First posted 2016-04-13 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hyperpolarised xenon (Other): evaluating the sensitivity of pulse sequences for 129Xe magnetic resonance imaging in the lungs, heart and brain and monitoring the transient changes in vital signs during and following the gas inhalation
  Interventions: Other: Hyperpolarised Xenon

INTERVENTIONS:
Other: Hyperpolarised Xenon — Hyperpolarised gas Magnetic resonance imaging (MRI) (3He and 129Xe) has enabled novel methods of in-vivo functional lung imaging that do not rely on the use of ionising radiation.

SUMMARY:
Hyperpolarised gas Magnetic resonance imaging (MRI) (Hyperpolorised 3He and 129Xe MRI) provides novel regional functional images of the lungs. Over the past 14 years researchers at Sheffield Teaching Hospitals NHS Foundation Trust and University of Sheffield have been developing and evaluating different MRI techniques to investigate different aspects of the lung function with both Hyperpolorised 3He and more recently 129Xe gas and have tested these new methods in volunteers with healthy and diseased lungs. This proposed study is to further test the sensitivity of MRI pulse sequences with inhaled 129Xe gas in volunteers. This protocol serves to evaluate the sensitivity of pulse sequences for 129Xe magnetic resonance imaging in the lungs and monitoring the transient changes in vital signs during and following the gas inhalation. This includes evaluation of pulse sequences to image xenon in the heart and brain as well as in the lungs of volunteers.

DETAILED DESCRIPTION:
The primary endpoints are to test the pulse sequences under development to image lung ventilation and perfusion, cardiac perfusion and brain uptake of xenon

The study will seek to test the given pulse sequence under investigation in a group of up to 40 volunteers.

To be eligible, each subject will have no contraindications to MRI scanning and will have signed the necessary volunteer consent forms.

The target recruitment number should provide sufficient data to determine the efficacy of the techniques under development.

Methods HP 129Xe MRI scans will be performed. MRI images will be acquired with the patients supine inside a 129Xe-capable MRI system, (1.5 Tesla GE, USA or 3.0 Tesla Philips, Netherlands), using dedicated transmit-receive radio-frequency coils.

129Xe is hyperpolarised on site to >50% polarisation using a Rubidium spin exchange polariser, and administered through a Tedlar bag. The 129Xe polarisation process has regulatory approval as an IMP for lung imaging from the MHRA (UK-MAIMP-29724). 129Xe will be manufactured as required for study volunteers. Manufactured 129Xe is held in a bag prior to administration to the study participant. Bags of manufactured gas will be labelled using labels approved by the MHRA. Drug accountability records will be held in the site file to document the administration of 129Xe to study participants. Hyperpolarised 129Xe will be prescribed to the participants prior to administration by a medically qualified study investigator using the study-specific prescription.

Subjects will be asked to go through several test runs of the inhalation procedure prior to imaging without actually starting to inhale the contents of the administration bag. The subject's heart rate and oxygen saturation will be monitored continuously during the studies using magnetic resonance compatible monitoring equipment.

ELIGIBILITY:
Inclusion Criteria:

* Any sex.
* Age greater than 18, less than 80.

NB: Participants will also be permitted to take part in study STH15080 (Eudract number 2009-010815-34, 'Development of new Magnetic resonance imaging (MRI) pulse sequences for probing lung function in volunteers with hyperpolarised 3He gas').

Exclusion Criteria:

* Contraindication to MRI.
* Resting oxygen saturation less than 90%.
* Known disease of the lungs, heart or brain.
* Pregnant.

Volunteer eligibility will be determined by completion of the study screening form not by physical examination or testing. Eligibility will be confirmed by a clinician upon review of the study screening form, prior to completing the study prescription for xenon dosing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of images 1 | Baseline
  signal to noise ratio,
Qualitative assessment of images 2 | Baseline
  spatial resolution
Qualitative assessment of images 3 | Baseline
  presence of artifacts

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffiths, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Academic Unit of Radiology, Univeristy of Sheffield, Sheffield, South Yorkshire, United Kingdom